CLINICAL TRIAL: NCT01592058
Title: Weight Change Among Users of Three Progestin-Only Methods of Contraception Over a 12-Month Time Period
Acronym: BMI
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201102211
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Weight Change
Keywords: weight change; contraception; birth control; progestin; progestin only; weight gain; depo; Depo Provera; DMPA; IUD; IUC; Mirena; Paragard; Implanon; implant
MeSH Terms: conditions — Body Weight Changes; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn whether women who use progestin-only methods of birth control such as the contraceptive implant (Implanon), the levonorgestral-releasing IUS (Mirena), or depot medroxyprogesterone acetate(DMPA) will experience weight change compared to women using the non-hormonal copper IUC (ParaGard).

The investigators primary hypothesis is that users of DMPA will gain excess weight and increase their BMI above the copper-IUC users; secondarily, the investigators will compare users' data in the LNG-IUC and ENG implant groups to the copper-IUC group.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in CHOICE between the ages of 18 and 45 who consented to future studies
* Chose levonorgestrel-releasing IUD, copper IUD, the implant, or DMPA as their CHOICE baseline method
* Has baseline height and weight data collected from the on-campus enrollment site
* Able to come back to the on-campus enrollment site for consent process and enrollment activities

Exclusion Criteria:

* Recent history of DMPA use before starting their baseline CHOICE method
* Used current method for less than 11 months or more than 12 months and three weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants already enrolled in the Contraceptive CHOICE Project will be offered participation during their 12-month follow up window if they had originally selected one of the four methods being studied during CHOICE enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline and 12 months
  Change in weight from baseline at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa E Madden, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: The Contraceptive CHOICE Project website - parent study for BMI — http://www.choiceproject.wustl.edu/